CLINICAL TRIAL: NCT01191866
Title: Intensive Individual and Familial Psychosocial Interventions in the Treatment of Children and Adolescents With Type 1 Diabetes Mellitus
Brief Title: Psychosocial Interventions in the Treatment of Youth With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr. Shira Shacham, Assaf Harofeh Pediatric Diabetes Clinic
Other Study IDs: 0406
Record Dates: First submitted 2010-08-29; First posted 2010-08-31 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; psychosocial; metabolic control; quality of life questionnaires; children; adolescents
MeSH Terms: conditions — Diabetes Mellitus | interventions — Psychosocial Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes mellitus: All children and adolescents with type 1 diabetes mellitus attending Assaf Harofeh Pediatric Diabetes Clinic
  Interventions: Behavioral: psychosocial intervention

INTERVENTIONS:
Behavioral: psychosocial intervention — The interventions will include an art therapist, a social worker and volunteer work under the supervision of a diabetes nurse. These therapies will be given to selected patients based on individual needs. We will use existing questionnaires in order to identify problematic areas and quantify quality of life

SUMMARY:
Primary Objective is to evaluate the influence of psychosocial interventions in the treatment of children and adolescents with type 1 diabetes mellitus by measuring the connection between these interventions to quality of life and to metabolic control. Secondary Objective is to provide an opportunity, through quality of life (QOL) questionnaires, for enhanced communication between the patient, family and diabetes care team and also an opportunity to resolve negative issues.

ELIGIBILITY:
Inclusion Criteria:

* All children and adolescents with type 1 diabetes mellitus attending Assaf Harofeh Pediatric Diabetes Clinic will be eligible for inclusion in the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children and adolescents with type 1 diabetes mellitus attending Assaf Harofeh Pediatric Diabetes Clinic will be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Pediatric Diabetes Clinic, Ẕerifin, Israel